CLINICAL TRIAL: NCT01420458
Title: A Randomized, Two-Period Crossover Study in Healthy Volunteers to Establish the Bioequivalence of Two Formulations of BG00012.
Brief Title: Study in Healthy Volunteers to Establish the BioEquivalence of Two Formulations of BG00012
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Biogen (Industry)
Responsible Party: Medical Director, Biogen Idec
Allocation: Randomized | Model: Crossover | Masking: None
Other Study IDs: 109HV107
Record Dates: First submitted 2011-08-11; First posted 2011-08-19 (Estimated); Last update posted 2011-11-04 (Estimated); Status verified 2011-11

CONDITIONS: Healthy Volunteers
Keywords: bioequivalence

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Drug: Experimental — Bioequivalence of two drug formulations

SUMMARY:
This is an open-label, single-center, 2 period crossover, PK profile study. Each subject will be randomized to 1 of 2 treatment sequences. Both treatment sequences will be enrolled concurrently.

DETAILED DESCRIPTION:
This is a study of healthy volunteers to demonstrate bioequivalence of two formulations of BG-00012 given in capsule form..

ELIGIBILITY:
Inclusion Criteria:

* Must give written and informed consent and any authorizations required by local law.
* Males and females 18 - 55 years old inclusive at time of consent.
* Must have a body mass index (BMI) between 19 kg/m2 and 30 kg/m2, inclusive

Exclusion Criteria:

* History of malignancy (subjects with basal cell carcinoma that has been completely excised prior to study entry remain eligible).
* Known history of or positive test result for Human Immunodeficiency Virus (HIV)
* History of severe allergic or anaphylactic reactions.
* History of any clinically significant cardiac, endocrinologic, hematologic, hepatic, immunologic,metabolic, urologic, pulmonary, neurologic, dermatologic, psychiatric and renal or other major disease, as determined by the Investigator.
* Clinically significant abnormal hematology or blood chemistry values, as determined by the Investigator, and any screening values for alanine aminotransferase (ALT) aspartate aminotransferase (AST) total bilirubin, or creatinine above the upper limit of normal, or an out of normal range screening value for white blood cells (WBC).
* Current enrollment in any other drug, biologic, or device study.

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 80 (Actual)
Dates: Start 2011-08; Primary Completion 2011-09 (Actual); Study Completion 2011-09 (Actual)

PRIMARY OUTCOMES:
Area under the plasma concentration curve as a measure of PK. | Participants will be followed during the duration of the study, 4 days. Samples taken at -15mins, 30 mins, 60 mins, 90 mins, 2 hrs, 3 hrs, 4 hrs, 5 hrs, 6 hrs, 7 hrs, 8 hrs, 10 hrs, 12 hrs

SECONDARY OUTCOMES:
The number of AEs in participants as a measure of safety and tolerability. | Participants will be followed during the time of study - an estimated four days

CONTACTS AND LOCATIONS:
Locations (1):
- Research Site, Minneapolis, Minnesota, United States